CLINICAL TRIAL: NCT04523285
Title: A Phase I, Open-label, Dose Escalation and Expansion Study to Evaluate the Tolerance, and Pharmacokinetics of TQB3728 Tablets
Brief Title: A Phase I Study of TQB728 Tablets on Tolerance and Pharmacokinetics
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3728-I-01
Record Dates: First submitted 2020-08-20; First posted 2020-08-21 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-08

CONDITIONS: Advanced Solid Tumor or Hematologic Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3728 tablets (Experimental): TQB3728 tablets administered orally, once a week in 28-day cycle.
  Interventions: Drug: TQB3728

INTERVENTIONS:
Drug: TQB3728 — TQB3728 tablets is a small molecule oral drug.

SUMMARY:
This is a open-label, phase I study to evaluate tolerance and pharmacokinetics of TQB3728 tablets in subjects with advanced solid tumor or hematologic tumor.

ELIGIBILITY:
Inclusion Criteria:

* 1.Understood and signed an informed consent form. 2.Histologically or cytologically confirmed advanced/metastatic or refractory solid tumor or lymphoma. No approved standard treatment regimen or ineffective or intolerant to standard treatment regimen.

  3.Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2; Life expectancy ≥12 weeks.

  4. Has at least one measurable lesion (solid tumors based on RECIST V1.1, lymphoma based on Lugano 2014).

  5.Adequate organ system function. 6.Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the first administration.

Exclusion Criteria:

* 1.Hypersensitivity to TQB3728 or its excipient. 2.Has received chemotherapy, radiotherapy, hormone therapy, immunotherapy, targeted therapy, biotherapy or any other antitumor therapy within 4 weeks before first administration.

  3.Has received allogeneic hematopoietic stem cell transplantation or organ transplantation, or received autologous hematopoietic stem cell transplantation within 12 weeks before administration.

  4.Has multiple factors affecting oral medication. 5.Has primary CNS lymphoma or CNS metastasis with untreated or uncontrolled symptoms.

  6.Pregnant or lactating women. 7.Has severe or uncontrolled systemic disease. 8.Has serious cardiovascular diseases. 9.Has neurological or mental disorders. 10.Has autoimmune disease or diseases requiring systemic hormones or immunosuppressive drugs.

  11.Has active viral infection. 12.The related toxicity of previous anti-tumor therapy has not recovered to CTCAE ≤ grade 1, except for hair loss.

  13. Has received major surgery within 4 weeks before the first administration. 14.Has participated in other clinical trials within 4 weeks before participating in this trial.

  15.According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Baseline up to 28 days
  MTD was defined as the dose in which more than 2 of up to 6 patients developed a DLT.

SECONDARY OUTCOMES:
Tmax | 30minutes pre-dose on day 1and day 8;1hour, 2hour, 3hour, 4hour, 6hour, 8hour, 24hour, 72hour post-dose on day 1 and day 8; 48hour, 96hour post-dose on day 1.
  To characterize the pharmacokinetics of TQB3728 by assessment of time to reach maximum plasma concentration.
Cmax | 30minutes pre-dose on day 1and day 8;1hour, 2hour, 3hour, 4hour, 6hour, 8hour, 24hour, 72hour post-dose on day 1 and day 8; 48hour, 96hour post-dose on day 1.
  Cmax is the maximum plasma concentration of TQB3738 or metabolite(s).
AUC0-t | 30minutes pre-dose on day 1and day 8; 1hour, 2hour, 3hour, 4hour, 6hour, 8hour, 24hour, 72hour post-dose on day 1 and day 8; 48hour, 96hour post-dose on day 1.
  To characterize the pharmacokinetics of TQB3728 by assessment of area under the plasma concentration time curve from zero to specific time or infinity.
Progression-free survival (PFS) | up to 48 weeks
  PFS defined as the time from first dose to the first documented progressive disease (PD) or death from any cause.
Overall response rate (ORR) | up to 48 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR).

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China